CLINICAL TRIAL: NCT07020416
Title: Transcutaneous Electrical Acustimulation in Automatic Synchronization With Breathing for Treating Functional Dyspepsia: A Phase I Feasibility Trial
Brief Title: AutoSTEA for Adults With Functional Dyspepsia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00000169
Record Dates: First submitted 2025-04-30; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with functional dyspepsia (Experimental): The treatment this arm will be administered is the AutoSTEA treatment, which consists of a band-like device that wraps around the rib cage. This device is connected to a microstimulator which is then connected to TENS pads. The band allows for the electrical impulses given to be synchronized with one's breathing.
  Interventions: Device: Transcutaneous electrical acustimulation in automatic synchronization with breathing

INTERVENTIONS:
Device: Transcutaneous electrical acustimulation in automatic synchronization with breathing — This intervention will be carried out via the AutoSTEA device.

SUMMARY:
The goal of this study is to assess how effective the AutoSTEA device is in treating functional dyspepsia (upper abdominal discomfort) in adults. It will also assess the safety and usability of the device. The main questions it aims to answer are:

* Does the AutoSTEA device ease dyspepsia symptoms?
* Is the AutoSTEA device safe and feasible for patients to use at their home?

Participants will:

* Use the device for half an hour every day for two weeks
* Have a phone check-in halfway through the trial
* Answer the daily and weekly questionnaires which consist of questions regarding symptoms, device usability, and adverse events experienced.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Must meet Rome IV criteria for functional dyspepsia

Exclusion Criteria:

* Patients with dyspepsia symptoms that have been fully resolved by antisecretory, antidepressant, or prokinetic therapy
* History of active NSAID use, unhealed esophagitis, unhealed ulcer disease, or other GI diseases that can explain their dyspepsia symptoms.
* History of upper GI surgeries and upper GI cancers, uncontrolled diabetes (type 1 and 2), severe psychiatric conditions, uncontrolled medical disorders, total knee replacement surgery, or above-the-knee amputation.
* Patients with H. pylori infection without confirmed eradication will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Determine the device safety when self-administered at home by patients | From enrollment to the end of treatment in two weeks
  Assess any adverse effects the device may have when used by patients in their home. This will be done using the device safety questionnaire. The safety questionnaire is to filled out weekly, with any adverse event that is experienced being reported. These adverse events (if applicable) will be rated in severity on a 0-5 scale, with 0 being the least severe and 5 being the most severe.
Evaluate device usability | From enrollment to the end of treatment in two weeks
  Assess how easy the device is for patients to use in their home. This will be done using the usability questionnaire. This questionnaire will be filled out daily and the user will rate on a 0-5 scale (with 0 being the worst and 5 being the best) how easy and comfortable the device was for them.
Assess symptom responses to treatment | From enrollment to the end of treatment in two weeks
  Assess how well a patient's dyspepsia symptoms respond to the treatment. This will be done via two questionnaires. One will be filled out weekly, where patients describe how much their dyspepsia symptoms have affected their daily lives. The scale for this will be 0-4, with 0 being no effect on their daily life and 5 being extreme effect on their daily lives. The second questionnaire will be filled out daily, and it describes the physical dyspepsia symptoms experienced by the patient in the last 24 hours. It is done on a scale from 0-10, with 0 meaning they have not experienced a symptom at all, and 10 being they have severely experienced a symptom.

SECONDARY OUTCOMES:
Assess a diverse participant pool, especially overweight/obese female patients | From enrollment to the end of treatment in two weeks
  Assess the response that patients have with a focus on those who are overweight/obese and female. This will be analyzed via the two dyspepsia symptom questionnaires that are mentioned in outcome 3.
Assess patient's compliance to AutoSTEA treatment | From enrollment to the end of treatment in two weeks
  Assess if patients followed through with the required usage of the device and treatment. This will be done via their own self-reporting to study staff of if they missed any treatment days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurin, MD, Principal Investigator — MetroHealth Medical Center
Locations (2):
- United States (2):
  - MetroHealth Medical Center - Main Campus, Cleveland, Ohio
  - MetroHealth Parma Medical Center, Parma, Ohio

IPD SHARING:
Plan to Share IPD: No
This data is preliminary data which we will use for IP protection and pattern application. We will keep the data confidential prior to future publication.

DOCUMENTS (2):
  • Study Protocol (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT07020416/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT07020416/SAP_001.pdf